CLINICAL TRIAL: NCT02042053
Title: Multimodality Imaging Assessment of Sipuleucel T Treatment and in Vivo Immune Response of Metastatic Castration Resistant Prostate Cancer Patients
Brief Title: PET/MR Assessment of Sipuleucel T Treatment for Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to PI leaving the institution
Sponsor: NYU Langone Health (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NYU S12-03902
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: imaging; diagnostic; castration resistant; metastatic prostate cancer; immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MR (Experimental): Patients treated with SipT (standard of care) undergo FDG-PET/MRI, NaF-PET/CT and blood drawing at 3 time points: baseline, Day 7 after the last SipT infusion, Week 10 after the last SipT infusion.
  Interventions: Device: PET/CT; Device: PET/MRI

INTERVENTIONS:
Device: PET/CT
Device: PET/MRI

SUMMARY:
This study intents to provide an initial evaluation of the utility of positron emission tomography and magnetic resonance (PET/MR) imaging measures for the prediction of immunological response to Sipuleucel T (SipT) therapy.

DETAILED DESCRIPTION:
Recent studies of treatments of prostate cancer through stimulation of adaptive immune response have indicated the linear measurements by computed tomography (CT) and nuclear scans used to assess tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) were inadequate and the value of progression-free survival (PFS) as a predictive surrogate endpoint of survival was lost.

The objective of this study is to provide an initial evaluation of the utility of PET/MR imaging measures for the prediction of immunological response to SipT therapy. Investigators expect to identify an"imaging-signature" of response to SipT based on changes in metabolism, perfusion, oxygenation and cellularity of metastasis and its correlation with immunological and clinical response. This approach will help elucidate the mechanism of activity and dynamics of immune antitumor responses to SipT in vivo and to identify new parameters of tumor response and predictive value than current RECIST and PFS standards.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years of age
* History of prostate cancer treated with androgen deprivation
* Serum Testosterone levels <50 ng/mL
* Established asymptomatic or minimally symptomatic metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status≤2
* Accept the terms of the imaging modalities and performance at pre-established time points as described in the protocol and consent
* Accept the terms for immune-monitoring blood drawing and performance at pre-established time points as described in the protocol and consent
* Patients that are on steroids (prednisone up to 10mg daily or hydrocortisone 20 mg daily) alone or in combination with Zytega or ketoconazole prior to enrollment are eligible
* Patients that are on steroids for an underlying chronic condition are eligible. (prednisone up to 10 mg daily, dexamethasone <2 mg daily or fludrocortisone 0.1 mg daily orally)

Exclusion Criteria:

* Chemotherapy or radiation therapy treatment within 21 days of Sipuleucel-T
* ECOG performance status >2
* Prior treatment with Sipuleucel-T
* Patients with a history of another primary malignancy within the last 2 years that was not curatively treated, excluding basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Active spinal cord compression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with imaging parameter change(s) among the patients with immunological response | up to 14 weeks
  NaF-PET/CT, FDG-PET/MRI, and blood drawing (for immunological response) are performed on patients at baseline, day 7 after the last SipT infusion, and week 10 after the last SipT infusion. The changes in SUV (standard uptake value) max on FDG-PET and NaF-PET, in MRI-ADC (apparent diffusion coefficient ) value, in MRI contrast enhancement, and in T2 lesion size will be measured.

SECONDARY OUTCOMES:
Percentage of patients with imaging parameter change(s) among the patients who respond per Response Evaluation Criteria In Solid Tumors (RECIST) | up to 14 weeks
  NaF-PET/CT, FDG-PET/MRI, and blood drawing (for immunological response) are performed on patients at baseline, day 7 after the last SipT infusion, and week 10 after the last SipT infusion. The changes in SUV max on FDG-PET and NaF-PET, in MRI-ADC value, in MRI contrast enhancement, and in T2 lesion size will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ferrari, MD, Principal Investigator — New York University Cancer Center
Locations (1):
- New York University Cancer Center, New York, New York, United States